CLINICAL TRIAL: NCT02648568
Title: Does Hypnosis Improve Severe Sleepwalking ?
Acronym: HYPNOSOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P130603; 2014-A00791-46 (Other: IDRCB)
Record Dates: First submitted 2015-12-15; First posted 2016-01-07 (Estimated); Last update posted 2017-12-08 (Actual); Status verified 2017-09

CONDITIONS: Sleepwalking
Keywords: Sleepwalking; sleep terrors; arousal disorders; F513 (CIM-10); F514 (CIM-10)
MeSH Terms: conditions — Somnambulism; Night Terrors | interventions — Hypnosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hypnosis plus relaxation (Active Comparator): Ericksonian hypnosis, based on sensations when awakening partially during N3 ; Jacobson relaxation, based on flexion and relaxation of muscles (serves here as a control procedure)
  Interventions: Behavioral: Hypnosis plus relaxation
- Relaxation (Active Comparator): Jacobson relaxation, based on flexion and relaxation of muscles (serves here as a control procedure)
  Interventions: Behavioral: Relaxation

INTERVENTIONS:
Behavioral: Hypnosis plus relaxation — The patient will have 20 min of Jacobson 's type relaxation, with sequential contraction and relaxation of limb muscles followed by an induction of hypnosis based on the preferential channel of each patient and, during trance, recommendation to assimilter the bed room and bed to a safe place
  Arms: Hypnosis plus relaxation
Behavioral: Relaxation — The patient will have 20 min of Jacobson 's type relaxation, with sequential contraction and relaxation of limb muscles
  Other Names: Jacobson type relaxation
  Arms: Relaxation

SUMMARY:
The aim of the study is to compare the benefit of two cognitive therapies in severe sleepwalking/ sleep terrors: relaxation vs. relaxation plus hypnosis. This is a monocentric, double-blind controlled study. 75 patients (aged more than 15 yo) with severe sleepwalking (defined as at least one epsidoe per week and at least two awakenings in stage N3 on video polysomngraphy) will be included. All patients will have a visit 1 for diagnosis including a medical interview, a video polysomnography, questionnaires on sleepwalking (PADSS and systematized interview), sleep quality (PSQI, MEQ) and sleepiness (Epworth scale) and suggestibility scale. 25 patients will be randomized to the relaxation group, 25 patients to the hypnosis plus relaxation group, while the 25 non-randomized patients will be non-treated controls. Randomized patients will receive the therapy on day 1, and be monitored during the subsequent night. They will have a weekly therapy for 4 additional sessions and be monitored again on Month 1, as well as they will complete the sleep and sleepwalking questionnaires. They will also complete the questionnaire by phone on Month 3. The non-randomized controls will complete the questionnaire on month 1, with no therapeutical intervention between Day 1 and Month 1. The main outcome will be the frequency of sleepwalking episodes, as assessed by the PADSS-B. Secondary outcomes include the changes in other subitems of teh PADSS, of the N3 awakenings in v-PSG between night 1 and Night 2 (short term effect) and Night 1 and Night 28 (long term effect), as well as changes in sleep quality and sleepiness scales. A comparison of spectral EEG, as well as respiration, eye movements, muscle tone and heart rate during rest, hypnosis trance, relaxation and sleepwalking episodes is also scheduled.

DETAILED DESCRIPTION:
Extended description of the protocol, including more technical information (as compared to the Brief Summary) if desired. Do not include the entire protocol; do not duplicate information recorded in other data elements, such as eligibility criteria or outcome measures

ELIGIBILITY:
Inclusion Criteria

1. >15 years old
2. French speaker
3. having signed the Informed consent form
4. Affiliated to National Health Insurance
5. Sleepwalking or sleep terrors (ICSD-3 criteria);
6. At least 2 awakenings from N3 on Night 1 videopolysomnography;
7. At least one episode per week.

Exclusion Criteria

1. < 15 years old
2. Patient under guardian ship
3. Patient unable to understand the protocol
4. Patient unable, from investigator's opinion, to comply to the procedures of the trial, including the ability to practice self-hypnosis.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Frequency of sleepwalking episodes as assessed by the PADSS-B | at one month (long term)
  PADSS-B questionnaire, including the frequency of sleepwalking/sleep terrors episodes as evaluated by the patients, from none(0) to (several par nights (6)

SECONDARY OUTCOMES:
Other subjective characteristics of sleepwalking/sleep terrors | At one and at three months
  total PADSS score
Objective measures of sleepwalking: number of N3 awakenings | Night 2 (8 hours) and at one month (long term)
  Number of N3 awakenings
Objective measures of sleepwalking :behaviors on videoPSG | Night 2 (8 hours) and at one month (long term)
  scale of behaviors on videopSG
% of sleep stages | Night 2 (8 hours) and at one month (long term)
  sleep stages (% of total sleep time)
total sleep time | Night 2 (8 hours) and at one month (long term)
  total sleep time in minute
sleep efficiency | Night 2 (8 hours) and at one month (long term)
  ratio between total sleep time and total sleep period
Spectral EEG (power) | At night 1 (8 hours)
  Spectral EEG analysis during hypnotic trance, rest, relaxation and N3 awakenings
Eye movements (number per minute) | At night 1 (8 hours)
  EOG during rest, hypnotic trance, relaxation, and N3 awakenings
Muscle tone (amplitude in microvolt) | At night 1 (8 hours)
  chin EMG during rest, hypnotic trance, relaxation, and N3 awakenings
Respiration (Rate of breathing per minute) | At night 1 (8 hours)
  Respiratory rate and amplitude via impedance belts during rest, hypnotic trance, relaxation, and N3 awakenings
Heart rate (beats per minutes) | At night 1 (8 hours)
  heart rate via ECG during rest, hypnotic trance, relaxation, and N3 awakenings
Frequency of sleepwalking episodes as assessed by the PADSS-B | at three months (very long term)
  PADSS-B questionnaire, including the frequency of sleepwalking/sleep terrors episodes as evaluated by the patients, from none(0) to (several par nights (6)
REM sleep without atonia | At night 1 (8 hours)
  Per % of tonic and phasic enhanced muscle tone during REM sleep

CONTACTS AND LOCATIONS:
Overall Officials: ARNULF Isabelle, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Groupe Hospitalier Pitié-Salpétrière, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barros A, Uguccioni G, Salkin-Goux V, Leu-Semenescu S, Dodet P, Arnulf I. Simple behavioral criteria for the diagnosis of disorders of arousal. J Clin Sleep Med. 2020 Jan 15;16(1):121-128. doi: 10.5664/jcsm.8136. Epub 2019 Dec 4. PMID 31957639
- [Derived] Dubessy AL, Leu-Semenescu S, Attali V, Maranci JB, Arnulf I. Sexsomnia: A Specialized Non-REM Parasomnia? Sleep. 2017 Feb 1;40(2). doi: 10.1093/sleep/zsw043. PMID 28364495